CLINICAL TRIAL: NCT00528840
Title: A Phase 3, Open-Label Study of the Safety and Efficacy of AA4500 in the Treatment of Subjects With Advanced Dupuytren's Disease
Brief Title: Safety and Efficacy Study of AA4500 (XIAFLEX™, Proposed Name) in the Treatment of Advanced Dupuytren's Disease
Acronym: JOINT-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-856
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2010-10-22 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Advanced Dupuytren's Disease
MeSH Terms: interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AA4500 0.58 mg (Experimental)
  Interventions: Biological: collagenase clostridium histolyticum

INTERVENTIONS:
Biological: collagenase clostridium histolyticum — Up to five injections of AA4500 into cord(s) of the affected hand(s). Each injection was separated by at least 30 days.
  Other Names: XIAFLEX®; AA4500

SUMMARY:
This was a Phase 3, 9-month, open-label study conducted in the United States. Subjects with a diagnosis of advanced Dupuytren's disease in a metacarpophalangeal (MP) or proximal interphalangeal (PIP) joint that resulted in a fixed flexion deformity of at least one finger, other than the thumb, that was at least 20° as measured by finger goniometry and was suitable for evaluation and injection were enrolled.

This study was designed to be part of the larger clinical program, for adult patients with Dupuytren's contracture with a palpable cord, where the data from 2 pivotal Placebo-Controlled studies (AUX-CC-857 (NCT00528606) and AUX-CC-859 (NCT00533273)) and 7 non-pivotal studies were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of advanced Dupuytren's disease, with a fixed flexion deformity of at least one finger, other than the thumb, that had a contracture at least 20°, but not greater than 100° for MP (80° for PIP) joints, caused by a palpable cord.
* Had a positive "table top test," defined as the inability to simultaneously place the affected finger(s) and palm flat against a table top.
* Were naïve to AA4500 treatment or had received one or two injections of AA4500 for the treatment of advanced Dupuytren's disease in Auxilium Studies AUX-CC-851, AUX-CC-853, or AUX-CC-855.
* Were judged to be in good health.

Exclusion Criteria:

* Had a chronic muscular, neurological, or neuromuscular disorder that affected the hands.
* Had received treatment for advanced Dupuytren's disease within 90 days of enrollment on the joint selected for the initial injection of AA4500, including surgery (fasciectomy or surgical fasciotomy), needle aponeurotomy/fasciotomy, or injection of verapamil and/or interferon.
* Had a known recent history of stroke, bleeding, a disease process that affected the hands, or other medical condition, which in the investigator's opinion, would make the subject unsuitable for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, Study Director — Endo Pharmaceuticals
Locations (14):
- United States (14):
  - Hope Research Institute, Phoenix, Arizona
  - Tucson Orthopedic Institute, P.C., Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - Southern Illinois Hand Center, S.C., Effingham, Illinois
  - Rockford Orthopedic Associates, Ltd., Rockford, Illinois
  - The Indiana Hand Center, Indianapolis, Indiana
  - Pri Via, Wichita, Kansas
  - St. Alexius Medical Center, Bismarck, North Dakota
  - David R. Mandel, Inc., Mayfield, Ohio
  - St. Vincent Medical Center, Portland, Oregon
  - Hamot Center for Clinical Research, Erie, Pennsylvania
  - Alpha Clinical Research, Clarksville, Tennessee
  - The Rheumatic Disease Clinic of Houston, Houston, Texas
  - Accurate Clincal Research, Houston, Texas

REFERENCES:
- See also: XIAFLEX Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/125338lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500 0.58 mg: collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
Period: Overall Study
Arm/Group | AA4500 0.58 mg
Started | 201
Completed | 168
Not Completed | 33
Not completed — Lost to Follow-up | 10
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 17
Not completed — Death | 2
Not completed — Administrative Reasons | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 164
Race/Ethnicity, Customized [Number; unit: participants]
  White | 201
Region of Enrollment [Number; unit: participants]
  United States | 201

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Contracture to 5° or Less
Description: The Primary Outcome Measure is the percentage of joints that were successfully treated where "successfully treated" was defined as reduction in contracture to within 0-5 degrees of normal within 30 days of injection
Time Frame: Within 30 days after the last injection
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Number; unit: percentage of joints
Units Other Than Participants: joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (joints) | 292
percentage of joints | 52.7

2. Secondary Outcome: Clinical Improvement After the Last Injection
Description: Clinical Improvement is defined as >=50% percent reduction from baseline in degree of contracture within 30 days after injection.
Time Frame: Baseline; within 30 days after last injection
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Number; unit: percent of joints
Units Other Than Participants: Number of joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (Number of joints) | 292
percent of joints | 71.6

3. Secondary Outcome: Percent Reduction From Baseline Contracture After the Last Injection
Description: Percent change in degree of contracture measured as 100*(baseline contracture -last available post-injection contracture)/baseline contracture)
Time Frame: Baseline, within 30 days after last injection
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Mean (Standard Deviation); unit: percentage of joints
Units Other Than Participants: joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (joints) | 292
percentage of joints | 66.8 (40.91)

4. Secondary Outcome: Change From Baseline Range of Motion After the Last Injection
Description: Change in degree of range of motion measured as last available post-injection range of motion - baseline range of motion.
Time Frame: Baseline, 30 days after last injection
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Number of Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (Number of Joints) | 292
degrees | 28.3 (20.15)

5. Secondary Outcome: Time to Reach Clinical Success
Description: Clinical success is defined as reduction in contracture to within 0-5 degrees of normal within 30 days of injection, displayed in post-injection timepoint categories.
Time Frame: First evaluation visit on which clinical success is achieved through the Day 30 evaluation
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Number; unit: percentage of joints
Units Other Than Participants: joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (joints) | 292
percentage of joints
  Injection 1, Day 1 | 9.6
  Injection 1, Day 7 | 16.4
  Injection 1, Day 30 | 16.1
  Injection 2, Day 0 | 0.0
  Injection 2, Day 1 | 2.4
  Injection 2, Day 7 | 2.4
  Injection 2, Day 30 | 3.1
  Injection 3, Day 0 | 0.0
  Injection 3, Day 1 | 0.7
  Injection 3, Day 7 | 1.0
  Injection 3, Day 30 | 0.7
  Injection 3, Day 90 | 0.3
  Did not reach clinical success | 47.3

6. Secondary Outcome: Clinical Success After the First Injection
Description: Clinical Success is defined as reduction in contracture to within 0-5 degrees of normal within 30 days of injection.
Time Frame: Within 30 days after first injection
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Number; unit: percentage of joints
Units Other Than Participants: joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (joints) | 292
percentage of joints | 42.5

7. Secondary Outcome: Clinical Improvement After the First Injection
Description: Clinical Improvement is defined as >=50% reduction from baseline in the degree of contracture within 30 days after the first injection
Time Frame: Baseline; within 30 days after first injection
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Number; unit: percentage of joints
Units Other Than Participants: joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (joints) | 292
percentage of joints | 64.4

8. Secondary Outcome: Percent Reduction From Baseline Contracture After the First Injection
Description: Percent change in degree of contracture is measured as 100* (baseline contracture- last available post-injection contracture)/baseline contracture.
Time Frame: Baseline; within 30 days after first injection
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Mean (Standard Deviation); unit: percentage of change
Units Other Than Participants: joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (joints) | 292
percentage of change | 60.4 (39.38)

9. Secondary Outcome: Change From Baseline Range of Motion After the First Injection
Description: Change in degree of range of motion measured as last available post-injection range of motion-baseline range of motion.
Time Frame: Baseline; within 30 days after first injection
Population: Intent to treat population (ITT) defined as all subjects who received at least one injection.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Joints
Arm/Group | AA4500 0.58 mg
Number analyzed (Participants) | 201
Number analyzed (Joints) | 292
degrees | 25.3 (19.52)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (non-SAEs) were collected from time of study drug administration, serious adverse events (SAEs) were collected from time subject signed ICF. Non-SAEs & SAEs were collected until 30 days after completion or discharge from study.
Description: This study was designed to be part of the larger clinical program, for adult patients with Dupuytren's contracture with a palpable cord, where the data from 2 pivotal Placebo-Controlled studies (AUX-CC-857 and AUX-CC-859) and 7 non-pivotal studies were evaluated.
Arm/Group | AA4500 0.58 mg
Serious Adverse Events (participants affected / at risk) | 11/201
Other Adverse Events (participants affected / at risk) | 197/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=201)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Finger amputation (Surgical and medical procedures) | 1 (1)
Intervertebral discitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rocky mountain spotted fever (Infections and infestations) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Thyroid gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=201)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Blood blister (Skin and subcutaneous tissue disorders) | 10 (11)
Contusion (Injury, poisoning and procedural complications) | 100 (174)
Ecchymosis (Skin and subcutaneous tissue disorders) | 43 (98)
Erythema (Skin and subcutaneous tissue disorders) | 12 (15)
Haematoma (Vascular disorders) | 12 (13)
Injection site haemorrhage (General disorders) | 109 (168)
Injection site pain (General disorders) | 116 (182)
Injection site pruritus (General disorders) | 19 (23)
Injection site swelling (General disorders) | 57 (98)
Oedema peripheral (General disorders) | 151 (431)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 (61)
Pruritus (Skin and subcutaneous tissue disorders) | 24 (35)
Skin laceration (Injury, poisoning and procedural complications) | 32 (36)
Swelling (General disorders) | 10 (13)
Tenderness (General disorders) | 48 (68)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Auxilium Pharmaceuticals, Inc. agreements may vary with individual investigators but will not prohibit any investigator from publishing. Auxilium supports the publication of results from all centers of a multicenter trial but requests that reports based on single site data not preceed the primary publication of the entire clinical trial.